CLINICAL TRIAL: NCT04836689
Title: Influence of Respiratory Rate Settings on CO2 Levels During Nasal Intermittent Positive Pressure Ventilation (NIPPV).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ori Hochwald , MD, Director, NICU, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMB-0490-20
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Ventilator Lung; Newborn
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Infants will be monitored by TcCO2 during three consecutive time periods of one hour each on a high and low rate of NIPPV, when in a stable condition. NIPPV rate will start high/low, changed to low/high and switched back to starting rate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 breaths per minutes (Other): Using NIPPV with rate of 30 for 1 hour. Measuring trans cutaneous CO2
  Interventions: Device: nasal intermittent positive pressure ventilation (NIPPV).
- 10 breaths per minute (Other): Using NIPPV with rate of 10 for 1 hour. Measuring trans cutaneous CO2
  Interventions: Device: nasal intermittent positive pressure ventilation (NIPPV).

INTERVENTIONS:
Device: nasal intermittent positive pressure ventilation (NIPPV). — NIPPV will be administered using Leoni (Heinen&Löwenstein, Bad Ems, Germany) and RAM cannula (Neotech, Valencia, CA).
  After initial setting and before routine blood gas testing, tcCO2 will be connected and calibrated. We will use SenTec digital monitor (SenTec AG, Therwil, Switzerland). Correlation/agreement between the tcCO2 and PCO2 will be assessed and documented in each infant.
  For Each infant we will get 2 set of data: Change in measurements when changing from 30 bpm to 10 bpm, and change in measurements when changing from 10 bpm to 30 bpm At the end of each hour, before rate change, we will document the following measurements:TcCO2, FiO2, saturation, the infant's respiratory rate (as measured in the monitor), number of apneas, bradycardia (heart rate<100 bpm), saturation<90% and>94% episodes (as measured in the monitor), 1-hour saturation histogram clasification.

SUMMARY:
Infants will be monitored by TcCO2 during three consecutive time periods of one hour each on a high and low rate of NIPPV, when in a stable condition. NIPPV rate will start high/low, changed to low/high and switched back to starting rate.

DETAILED DESCRIPTION:
This will be a prospective, crossover observational study that will be performed at Rambam NICU.

Infants will be monitored by TcCO2 during three consecutive time periods of one hour each on a high and low rate of NIPPV, when in a stable condition.

NIPPV rate will start high/low, changed to low/high and switched back to starting rate.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 240 to 336.
* At least 6 hours of stabilized NIPPV settings, i.e. minor changes in settings (FiO2 ≤0.10, PIP≤ 2.0 cmH2O, RR≤ 5 brm).
* At least 6 hours of stabilized tcCO2, i.e. ≤5 mmHg variation.
* At least 6 hours from surfactant administration.
* Parental consent

Exclusion Criteria:

* If NIPPV set rate is 10 bpm and tcCO2 related pCO2 is<40mmHg.
* If NIPPV set rate is 30 bpm and tcCO2 related pCO2 is>60mmHg.
* Unstable infants due to acute conditions (sepsis. IVH), or congenital malformations.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Trans cutaneous CO2 (TCCO2) | During the 3 hours of the study
  Trans cutaneous CO2

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hochwald O, Borenstein-Levin L, Dinur G, Jubran H, Littner Y, Breuer M, Kugelman A. The effect of changing respiratory rate settings on CO2 levels during nasal intermittent positive pressure ventilation (NIPPV) in premature infants. J Perinatol. 2023 Mar;43(3):305-310. doi: 10.1038/s41372-023-01614-7. Epub 2023 Feb 9. PMID 36759706